CLINICAL TRIAL: NCT05350150
Title: Non-invasive Vagus Nerve Stimulation in Patients Undergoing Electrophysiological Study (VNS-EPS)
Brief Title: Non-invasive Vagus Nerve Stimulation in Patients Undergoing Electrophysiological Study
Acronym: VNS-EPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-1109
Record Dates: First submitted 2022-04-01; First posted 2022-04-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Auricular Vagal Nerve Stimulation (Experimental): Patients will undergo a standard EPS with 4 catheters. Following the standard EPS, patients will be hooked up a Parasym device to provide transcutaneous electrical stimulation to the auricular branch of the vagus nerve, EPS will be repeated.
  Interventions: Device: Auricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Auricular Vagal Nerve Stimulation — The Parasym device will be placed on the patient's left tragus to provide transcutaneous electrical stimulation to the auricular branch of the vagus nerve.

SUMMARY:
The Non-invasive Vagus Nerve Stimulation in Patients Undergoing Electrophysiological Study is a single center, pilot, prospective study that aims at evaluating the effects of auricular vagus nerve stimulation (aVNS) on the human cardiac conduction system.

DETAILED DESCRIPTION:
The Non-invasive Vagus Nerve Stimulation in Patients Undergoing Electrophysiological Study is a single center, pilot, prospective study that aims at evaluating the effects of auricular vagus nerve stimulation (aVNS) on the human cardiac conduction system. In this study, we will enroll 10 healthy individuals presenting to the electrophysiology laboratory for an electrophysiological study (EPS). Patients will undergo a standard EPS with 4 catheters (coronary sinus catheter, His catheter, right ventricular catheter, and right atrial catheter). Following the standard EPS, patients will be hooked up a Parasym device to provide transcutaneous electrical stimulation to the auricular branch of the vagus nerve.

ELIGIBILITY:
Inclusion Criteria:

* Primary indication for EPS for the evaluation of cardiac conduction system or supraventricular tachycardia.

Exclusion Criteria:

* Previous EPS with ablation
* Previous failed ablation
* Known conduction system disease, right or left bundle branch block on EKG
* Pregnant women
* History of postural orthostatic tachycardia syndrome
* Patients who have had prior cervical vagotomy
* Patients with skin on the tragus that is broken or cracked
* Patients with a history of baseline cardiac disease or atherosclerotic cardiovascular disease, including congestive heart failure (CHF), known severe coronary artery disease or recent myocardial infarction (within 5 years) and patients diagnosed with narrowing of the arteries (carotid atherosclerosis)
* Patients with an active implantable medical device, such as a cardiac pacemaker, hearing aid implant, or any implanted metallic, implanted vagus nerve stimulator or electronic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Sinus Cycle Length | Pre procedure/procedure
  Sinus cycle length (msec)
Change in A-H Interval | Pre procedure/procedure
  A-H Interval (msec)
Change in H-V Interval | Pre procedure/procedure
  H-V interval (msec)
Change in QRS Duration | Pre procedure/procedure
  QRS Duration (msec)
Change in QT Duration | Pre procedure/procedure
  QT Duration (msec)
Change in Sinus Node Recovery Time | Pre procedure/procedure
  Sinus Node Recovery Time (msec)
Change in AV Node Wenckebach Cycle Length | Pre procedure/procedure
  AV Node Wenckebach Cycle Length (msec)
Change in AV Node Effective Refractory Period | Pre procedure/procedure
  AV Node Effective Refractory Period (ERP) (msec)
Change in Atrial Effective Refractory Period | Pre procedure/procedure
  Atrial Effective Refractory Period ERP (msec)
Change in Right Ventricular Effective Refractory Period ERP | Pre procedure/procedure
  Right Ventricular Effective Refractory Period ERP (msec)
Change in retrograde block cycle length | Pre procedure/procedure
  Retrograde Block Cycle Length (msec)
Change in Accessory Pathway Anterograde Effective Refractory Period ERP | Pre procedure/procedure
  Accessory Pathway Anterograde Effective Refractory Period (msec)
Change in Accessory Pathway Retrograde Effective Refractory Period ERP | Pre procedure/procedure
  Accessory Pathway Anterograde Effective Refractory Period (msec)
Supraventricular Tachycardia induction | Pre procedure/procedure
  Supraventricular Tachycardia induction
Supraventricular Tachycardia Termination | Pre procedure/procedure
  Supraventricular Tachycardia Termination

CONTACTS AND LOCATIONS:
Overall Officials: Stavros E Mountantonakis, MD, Principal Investigator — Northwell Health
Locations (1):
- Kristie Coleman, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stavrakis S, Stoner JA, Humphrey MB, Morris L, Filiberti A, Reynolds JC, Elkholey K, Javed I, Twidale N, Riha P, Varahan S, Scherlag BJ, Jackman WM, Dasari TW, Po SS. TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial. JACC Clin Electrophysiol. 2020 Mar;6(3):282-291. doi: 10.1016/j.jacep.2019.11.008. Epub 2020 Jan 29. PMID 32192678
- [Background] Stavrakis S, Humphrey MB, Scherlag BJ, Hu Y, Jackman WM, Nakagawa H, Lockwood D, Lazzara R, Po SS. Low-level transcutaneous electrical vagus nerve stimulation suppresses atrial fibrillation. J Am Coll Cardiol. 2015 Mar 10;65(9):867-75. doi: 10.1016/j.jacc.2014.12.026. PMID 25744003
- [Background] Stavrakis S, Elkholey K, Morris L, Niewiadomska M, Asad ZUA, Humphrey MB. Neuromodulation of Inflammation to Treat Heart Failure With Preserved Ejection Fraction: A Pilot Randomized Clinical Trial. J Am Heart Assoc. 2022 Feb;11(3):e023582. doi: 10.1161/JAHA.121.023582. Epub 2022 Jan 13. PMID 35023349